CLINICAL TRIAL: NCT04329234
Title: Korean Heart Failure Registry Ⅲ of Korean Society of Heart Failure
Brief Title: Korean Heart Failure Registry III
Acronym: KorHF-III
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Korean Society of Heart Failure (Unknown)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Other Study IDs: KorHF-III
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute heart failure: Patients with acute heart failure

SUMMARY:
KorHF III is a multi-center, nationwide, prospective registry of the Korean Society of Heart Failure, which enrolls patients with acute heart failure in Korea.

The aim of this registry is to analyze the etiology, treatment, treatment, and prognosis to develop strategies for managing acute heart failure.

ELIGIBILITY:
All consecutive hospitalized adult heart failure patients who fulfill one of 1-3 and 4

Inclusion Criteria:

1. Symptoms of heart failure
2. Signs of heart failure
3. Lung congestion in Chest-x-ray
4. Objective finding of structural and/or functional disorder of the heart or elevated natriuretic peptide levels

Exclusion Criteria:

1. Patients younger than 18 years old
2. Patients who do no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 5 years
  In-hospital mortality
Post-discharge mortality | 5 years
  Post-discharge mortality
Post-discharge re-hospitalization | 5 years
  Post-discharge re-hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yoon M, Kim EJ, Han SW, Park SM, Kim IC, Cho MC, Ahn HS, Shin MS, Hwang SJ, Jeong JO, Yang DH, Kim JJ, Choi JO, Cho HJ, Yoo BS, Kang SM, Choi DJ. The Third Nationwide Korean Heart Failure III Registry (KorHF III): The Study Design Paper. Int J Heart Fail. 2024 Apr 1;6(2):70-75. doi: 10.36628/ijhf.2024.0001. eCollection 2024 Apr. PMID 38694931